CLINICAL TRIAL: NCT02155179
Title: Embryo Kinetics and Sperm Quality. Depends on the Sperm Quality the Embryo Cleavage Rate?
Brief Title: Sperm Pathology Samples and Morphokinetics
Status: Completed | Type: Observational
Sponsor: IVI Madrid (Other)
Responsible Party: Sponsor
Other Study IDs: semen-esd
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Cylinical Embryo; Oligospermia
MeSH Terms: conditions — Oligospermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Good prognosis: Sperm samples >15mill/ml >30% progresive sperms
- bad prognosis: Sperm samples <5mill/ml <5% progresive sperms

SUMMARY:
The embryo kinetics may be a new prognostic factor for choosing the embryos with the highest implantation potential. In order to identify the factors that may affect the rate of embryo cleavage, there are many studies about morphokinetics and culture medium, oxygen tension, oocyte quality or type of medication used for ovarian stimulation. However there are no published data with respect to the influence of semen quality in the embryo kinetic.

In this study The investigators propose that the sperm quality may has influence in the embryo division.

ELIGIBILITY:
Inclusion Criteria:

* Sperm samples with more than 15 mill/ml of sperms, more than 40% of mobile sperms
* Sperm samples with less than 5 mill/ml of sperms, less than 10% of mobile sperms

Exclusion Criteria:

* sperm samples between 5 to 15 mil/ml of sperms and between 10% to 40% of mobile sperms

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sperms samples of assisted reproduction treatments
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2014-08; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
embryo division in 2, 3, 4, 5, 6, 7, 8, cells and blastocyst formation | between day 0 and day 5 of development
  Exact time of cell cleavages

CONTACTS AND LOCATIONS:
Overall Officials: david agudo, PhD, Principal Investigator — lab coordinator
Locations (2):
- Spain (2):
  - IVI MAdrid, Madrid
  - Madrid